CLINICAL TRIAL: NCT03619044
Title: The Use of FES-PET Imaging as a Tool to Detect a Possible Reversion of Estrogen Receptor (ER)-α Status in Patients With Metastatic Breast Cancer HER2 + and ERα Neg Treated With Trastuzumab + Pertuzumab + Taxane.
Acronym: REVER
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment rate
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18 SEIN 08
Record Dates: First submitted 2018-08-01; First posted 2018-08-07 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: HER2-positive Breast Cancer
Keywords: Metastatic breast cancer; FES-PET; HER2-positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with metastatic breast cancer (Other): Patients with metastatic breast cancer treated with trastuzumab + pertuzumab + taxane in the metastatic first line.
  Interventions: Other: 2 FES-PET Imaging will be performed:

INTERVENTIONS:
Other: 2 FES-PET Imaging will be performed: — * before treatment initiation
  * before treatment cycle 3 initiation

SUMMARY:
This is an exploratory, prospective and multicentric study aiming to highlight by FES-PET imaging that an anti-HER2 treatment by trastuzumab + pertuzumab can reverse the ERα status in patients with metastatic breast cancer HER2 + and ERα neg.

For each included patient, 2 FES-PET Imaging will be performed for the study (before cancer treatment initiation and before the cycle 3 of treatment) at the IUCT-O center (Institut Universitaire du Cancer de Toulouse).

Treatment (trastuzumab + pertuzumab + taxane) will be administered according to the current recommendations in each participant center.

Patients will be followed during the 3 cycles of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Patient with metastatic breast cancer HER2 + (IHC+++ and/or HER2 amplification in ISH according to ASCO recommendations), ERα neg (0% in IHC) and Progesterone Receptor neg (0% in IHC).
3. Patient eligible according to the investigator for a treatment with trastuzumab + pertuzumab + taxane in the metastatic first line.
4. Available biopsy of a tumor lesion (archived material) or biopsiable tumor lesion for study (primitive tumor or metastasis other than bone).
5. OMS ≤ 2.
6. For non-menopausal patients, use of an effective contraceptive method at entry into the study and for the duration of the study.
7. Patient affiliated to a Social Health Insurance in France.
8. Patient must provide written informed consent prior to any study specific procedures.

Exclusion Criteria:

1. Any previous treatment for metastatic disease.
2. Prior adjuvant treatment with anti-HER2 antibodies taken within 6 months.
3. Patient with isolated hepatic metastasis.
4. Patient with hemostasis disorders.
5. Unbalanced Diabetes.
6. Patient with usual formal contraindication to PET/TDM Imaging.
7. Patient who has already started trastuzumab + pertuzumab + taxane treatment.
8. Pregnant or breastfeeding women.
9. Any psychological, familial, geographical or sociological condition which does not allow to respect the medical follow-up and/or compliance to study procedure.
10. Patient protected by law.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-07-09 (Actual)

PRIMARY OUTCOMES:
The rate of patients with conversion of FES negative lesions in FES positive lesions. | Cycle 3 Day 1 for each patient.

SECONDARY OUTCOMES:
The rate of patients with FES positive lesions before treatment. | Cycle 4 Day 1 for each patient.
The adverse events due to FES-PET imaging evaluated by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03. | Cycle 4 Day 1 for each patient.

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Clinique Claude Bernard, Albi
  - Centre Hospitalier Auch, Auch
  - Clinique Capio La Croix Du Sud, Quint-Fonsegrives
  - Centre Hospitalier de Rodez, Rodez
  - IUCT-O, Toulouse
  - Clinique Pasteur, Toulouse